CLINICAL TRIAL: NCT05773469
Title: Energy Balance in Extreme Environments: Metabolic Adaptation to Energy Expenditure and Finding the EI Limit
Brief Title: Energy Balance in Extreme Environments: Finding the EI Limit
Acronym: StOMPE
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 595711
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Energy Expenditure; Atrophy, Muscular; Energy Intake
Keywords: polar; ultra endurance; doubly labelled water; energy expenditure; energy intake; limit
MeSH Terms: conditions — Muscular Atrophy | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exercise — Ski traverse of Greenland polar Icecap
Other: Nutrition — Maximising energy intake by consuming over the theoretical 2.4 x RMR

SUMMARY:
This project is feasibility study looking at extreme exercise and possible diet intervention study to counter muscle and weight loss during a 2 person Greenland Ski Traverse in April 2023. By increasing energy intake to above the currently theoretical capacity (2.5 x RMR) the aim is to test a method to find out if there is a maximum to energy intake and whether energy deficit can be minimised; weight loss attenuated, and whether muscle can be preserved. If not, what are the likely adaptive mechanisms and use this to inform future work on dietary interventions

DETAILED DESCRIPTION:
Prolonged endurance events provide a unique opportunity to study the physiological limits of human performance. When nutrition is adequate, maintaining weight is directly related to energy expenditure. In extreme environments however, such as ocean rowing, the investigators have shown that rowers lost 10% weight, had a high energy expenditure (5,000kcal/d or 3.1 x basal metabolic rate) which was not met by energy intake (EI). Even in the presence of over ~5000kcal food per day, rowers chose to eat only ~3800kcal/d (2.4 x RMR) and lost weight, rather than eat more. It is also rare, outside of elite performance, that EI is above 2.5 x RMR and is suggestive of some sort of regulatory mechanism. Previous work has shown that high energy expenditures (EE) are not sustainable over long periods and that EE decreases with duration, plateauing at around 2.5 x RMR. This is in attempt to balance energy requirements in order to minimise body mass loss and increase chances of survival. Using data from the previous PhD study in ocean rowers (Holsgrove-West., 1st PhD study), and extrapolating data from the studies used to model TEE and duration, and overfeeding studies, voluntary energy intake calculated from body mass loss were consistently around 2.4 x RMR, suggesting a possible numerical value to the limit of EI. This has not been measured experimentally. If the theory of maximal EI is true, any intake above the maximum [2.4 x RMR] cannot be used for energy and would be excreted. Any BM loss would therefore reflect difference between EE and the maximal EI, not the actual EI. To investigate the EI limit therefore requires simultaneous measurements of EE, EI and body mass changes whilst ensuring EI above the theoretical maximum.In the presence of energy deficit and body mass loss, ocean rowers demonstrated an adaptive response by selectively maintaining or losing muscle. Loaded muscles were preserved whilst unloaded muscles atrophied. An obvious countermeasure could be to load the muscles that wasted, but to what expense? With finite energy intake, and greater demand from the muscle mass, other components of EE such as RMR, NEAT or exercise component may compensate, or endure a greater body mass loss. This interaction warrants further investigation. Logistically it is difficult to ask rowers to exercise mid-race, and compliance would be unknown. An expedition that involves greater muscle involvement and high EE is needed. Trekking across Greenland provides the high EE environment without the lower limb disuse. In addition, due to logistical reasons of sample storage in ocean rowing, energy expenditure and intake were collected only in the final week of the row, and energy balance did not match with body mass loss. This would indicate a different energy deficit and different energy expenditure or intake earlier on in the row. These initial acute changes are unknown and possibly responsible for the large weight loss seen by the end of the row. This project will attempt to fill that gap and measure these initial changes by measuring daily EI and EE.EI is rarely measured alongside EE and body mass loss and instead inferred from EE. This study aims to establish whether this maximal EI exists, by directly measuring both components of energy balance and how the body compensates with changes in the components of EE.

ELIGIBILITY:
Inclusion Criteria:

*Partaking in ski traverse across Greenland April - May 2023

Exclusion Criteria:

* No neurological, neuromuscular, or musculoskeletal disorders that could impair the quality of the muscle. eg. CP, muscular dystrophy or SCI
* Not pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 2 persons undertaking a ski traverse across Greenland April - May 2023. 1 male and 1 female
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-11-26 (Actual)

PRIMARY OUTCOMES:
body mass loss | 4 weeks
  total amount of weight lost

SECONDARY OUTCOMES:
muscle loss | 4 weeks
  muscle thickness loss in upper, lower limbs and trunk
energy deficit | 4 weeks
  total energy deficit calculated from energy expenditure and energy intake as well as from body mass loss

CONTACTS AND LOCATIONS:
Overall Officials: Francis Stephens, Principal Investigator — University of Exeter
Locations (1):
- University, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data can be made available only to those listed on the collaborators list. There will be consent gained for sharing on anonymised data only.